CLINICAL TRIAL: NCT00925080
Title: Pivotal Study of the Intravenous Blood Glucose (IVBG) System, In-Clinic Setting
Status: Completed | Type: Observational
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Andrew K. Balo / SVP, Clinical and Regulatory Affairs, and Quality Assurance, DexCom, Inc.
Other Study IDs: PTL-900193, Rev01
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Device: IVBG

INTERVENTIONS:
Device: IVBG — Venous blood glucose measurement every 7.5 minutes for 72-hours

SUMMARY:
The purpose of this study is to evaluate safety and accuracy of the IVBG System (the "System") when used to track blood glucose in insulin treated subjects with diabetes mellitus in an in-clinic setting for up to 72 hours (per subject). Reference blood glucose measurements will be collected across the entire reportable range of the System (e.g., 40 400 mg/dL) with adequate sampling at the upper and lower ends of this range. IVBG System accuracy will primarily be assessed relative to ISO 15197 criteria (i.e., within ±15 mg/dL at YSI glucose levels < 75 mg/dL, and within ±20% at YSI glucose levels >75 mg/dL).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Willing to participate in one 72-hour in-clinic session during which up to 72 venous blood samples drawn for YSI measurement of glucose concentration (maximum sampling frequency of 4 per hour), a fingerstick blood glucose measurement will also be performed at the time of each YSI blood draw;
3. If instructed, be willing not to perform any activities that would result in submersion of the Sensor/Potentiostat in water or willing to wear a waterproof covering when submerging the Sensor/Potentiostat;
4. Have been diagnosed with insulin-requiring diabetes mellitus and are on multiple daily injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII) insulin therapy;
5. Able to speak, read, and write English.

Exclusion Criteria:

1. Have skin conditions or existing (or planned) medical instrumentation and/or dressings that preclude wearing the IVBG Sensor (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis, or surgical dressings at the proposed wear site);
2. Are pregnant (as demonstrated by a positive pregnancy test within 72-hours of device insertion);
3. Have a contraindication to placement of a dedicated peripheral IV line;
4. Have a known history of heparin-induced thrombocytopenia;
5. Current participation in another investigational study protocol (if a subject has recently completed participation in another drug study, the subject must have completed that study at least 30 days prior to being enrolled in this study);
6. Have any condition that, in the opinion of the Investigator, would interfere with their participation in the trial or pose an excessive risk to study staff handling venous blood samples (e.g., known history of hepatitis B or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with insulin-requiring diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
IVBG System accuracy will primarily be assessed relative to ISO 15197 criteria (i.e., within ±15 mg/dL at YSI glucose levels < 75 mg/dL, and within ±20% at YSI glucose levels >75 mg/dL). | 72-hours

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Profil Institute for Clinical Research, Chula Vista, California
  - Advanced Metabolic Care + Research, Escondido, California
  - Diabetes and Glandular Disease Research Associates, Inc., San Antonio, Texas